CLINICAL TRIAL: NCT00238862
Title: Efficacy of Amniotic Membrane Transplantation and Autologous Serum in Treatment of Persistent Epithelial Defects
Brief Title: Treatment of PED With AMT and Autologous Serum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP0511-P
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Corneal Epithelial Defect
Keywords: Diabetes; Corneal transplant; Neurotrophic keratitis; Post-bacterial keratitis; Metaherpetic keratitis
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Amniotic membrane transplantation
Drug: Autologous serum/BSS 20%

SUMMARY:
Patients with persistent corneal epithelial defects who have not responded to conventional therapy will be randomized to treatment with either amniotic membrane transplantation or autologous serum 20%. Outcome measures will be (1) presence or absence of complete re-epithelialization within 28 days and (2) retention of intact epithelium for at least 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Corneal epithelial defect of more than 14 days that has not responded to conventional therapy

Exclusion Criteria:

* Under age 18
* Pregnant/lactating females
* Patients with hemoglobin levels < 12 mg/ml
* Patients with limbal stem cell deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2005-10; Study Completion 2006-09

PRIMARY OUTCOMES:
Corneal re-epithelialization (= initial success)
Persistent corneal re-epithelialization (= lasting success)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Wagoner, MD, Principal Investigator — King Khaled Eye Specialist Hospital
Locations (1):
- King Khaled Eye Specialist Hospital, Riyadh, Saudi Arabia